CLINICAL TRIAL: NCT05863910
Title: Real World Evidence on the Use of Medical Cannabis in Pediatrics: A Prospective Observational Study
Brief Title: Real World Evidence on the Use of Medical Cannabis in Pediatrics
Acronym: CAN-RWE
Status: Recruiting | Type: Observational
Sponsor: University of Manitoba (Other)
Collaborators: The Canadian Collaborative for Childhood Cannabinoid Therapeutics (Unknown); Canadian Cancer Society (CCS) (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: CAN-RWE
Record Dates: First submitted 2023-02-13; First posted 2023-05-18 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Cancer; Epilepsy; Neurodevelopmental Disorders
Keywords: cannabinoids; cannabis; pediatrics
MeSH Terms: conditions — Neoplasms; Epilepsy; Neurodevelopmental Disorders; Marijuana Abuse | interventions — Medical Marijuana

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Epilepsy Cohort: For children with epilepsy, the following tools will be added for data collection at each time point:
  * Side effects: Pediatric Epilepsy Side Effects Questionnaire [PESQ]
  * Seizure frequency/severity: Seizure Diary Data Questionnaire
  Interventions: Drug: Medical Cannabis
- Cancer Cohort: For children with cancer, the following tools will be added for data collection at each time point:
  * Cancer symptom burden: Symptom Screening in Pediatrics Tool [SSPedi]
  * Cachexia: Pediatric Functional Assessment of Anorexia/ Cachexia Treatment [peds-FAACT]
  Interventions: Drug: Medical Cannabis
- General Pediatrics Cohort: There are no specific outcome scales added for this cohort.
  Interventions: Drug: Medical Cannabis

INTERVENTIONS:
Drug: Medical Cannabis — Any cannabis product that is available to participants through the Medical Cannabis Access Program is eligible to be included in this study.

SUMMARY:
CAN-RWE is an observational study that is following 500 children who have authorizations for medical cannabis for two years from across Canada.

DETAILED DESCRIPTION:
Pediatric patients (3 to 17 years) using medical cannabis (MC) for pain, sleep, mood, behaviour, seizures, treatment of cancer, or to manage symptoms related to cancer or cancer-treatment are eligible to join this 24-month study if they have a valid MC authorization.

Following screening, eligible participants will be contacted by the study coordinator. Following informed consent, study participants will record complete outcome measures on pain, sleep, mood (anxiety, depression and positive affect), behaviour, as well as report their cannabis use and indication-specific outcomes as applicable at 3, 6, 12, and 18 weeks, as well as 6, 12, 18 and 24-months.

ELIGIBILITY:
Inclusion Criteria:

* 3 to 17 years
* have a medical document provided by a prescribing health care practitioner (i.e. physician, nurse practitioner, etc.) for the use of medical cannabis
* medical cannabis is authorized for pain, sleep, mood, behaviour, seizures, cancer or cancer-treatment related symptom management
* ability to respond to electronic questionnaires in English

Exclusion Criteria:

* individuals using cannabis for medical purposes without a medical cannabis authorization from a health care provider
* those only using cannabis recreationally

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Population includes children (3 to 17 years) who are cannabis-naïve or experienced with a medical document provided by a prescribing health care practitioner (i.e. physician, nurse practitioner, etc.) for the use o medical cannabis primarily for pain, sleep, mood, behaviour, seizures, cancer or cancer-treatment related symptom management.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Patterns of cannabis use (caregiver-reported) | baseline to 24-months
  Describe patterns of cannabis use are described using a standard data collection form including dose and product type completed by caregivers at baseline, 3, 6, 12, and 18-weeks and 6, 12, 18 and 24-months

SECONDARY OUTCOMES:
Effectiveness in seizure cohort - seizure frequency | baseline to 24-months
  Longitudinal assessment for benefit signals in epilepsy seizure frequency/severity measure by a seizure diary
Effectiveness in seizure cohort - QOLCE | baseline to 24-months
  Longitudinal assessment for benefit signals including epilepsy related side effects measured using QOLCE
Effectiveness in oncology cohort - symptom burden | baseline to 24-months
  Longitudinal assessment for benefit signals in caregiver reported changes in symptom burden assessed using mini-SSPEDI (under 8 yr) and SSPEDI scales
Effectiveness in oncology cohort - cachexia | baseline to 24-months
  Longitudinal assessment of cachexia using Peds-FAACT
Adverse events | baseline to 24-months
  Cannabis-related adverse events and serious adverse events reported by caregivers using a standard AE data collection tool and categorized according to CTCAE v5.0 at baseline, 3, 6, 12, and 18-weeks and 6, 12, 18 and 24-months
Family related quality of life | baseline to 24-months
  Longitudinal assessment of cachexia using PedsQL
Changes in mood - anxiety | baseline to 24-months
  PROMIS short form scales for pediatric anxiety symptoms 8a v2.0
Changes in mood - depression | baseline to 24-months
  PROMIS short form scales for pediatric depression symptoms 8a v2.0
Changes in mood - positive affect | baseline to 24-months
  PROMIS short form pediatric positive affect scale 8a v2.0
Changes in sleep related impairment | baseline to 24-months
  PROMIS short form pediatric sleep related impairment scale 8a v2.0
Changes in pain interference | baseline to 24-months
  PROMIS short form pediatric pain interference scale 8a v2.0
Parental overall impression of behaviour | baseline-24months
  Parents/Caregivers will be asked to report on if their childs behaviour has improved or worsened and will have an open-ended text box to describe anything they want to tell us about changes in their child's behaviour.

CONTACTS AND LOCATIONS:
Overall Officials: Sapna Oberoi, MD, Principal Investigator — University of Manitoba; Taylor Lougheed, MD, Principal Investigator — Northern Ontario School of Medicine; Evan Lewis, MD, Principal Investigator — Neurology Centre of Toronto
Locations (1):
- U Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Undecided
summary level data will be available upon reasonable request with appropriate approval and oversight of a research ethics board.

REFERENCES:
- See also: For more information on our research team visit our website. — http://www.medcannkids.ca